CLINICAL TRIAL: NCT04853654
Title: Investigation of the Effects of Selective Exercise Training on Muscle Architecture, Balance, Function and Fatigue in Multiple Sclerosis
Brief Title: Investigation of the Effects of Selective Exercise Training in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanko University (Other)
Responsible Party: Principal Investigator, zekiye ipek katırcı kırmacı, assistant professor, Sanko University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ipekkirmaci
Record Dates: First submitted 2021-04-11; First posted 2021-04-21 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Multiple Sclerosis; Exercise
Keywords: multiple sclerosis; muscle architecture; Eccentric Exercise; Concentric Exercise
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Selective training (Experimental): selective training on lower extremity for 3 days/week
  Interventions: Other: exercise
- Downhill walking (Experimental): downhill walking training on the treadmill for 2 days/week
  Interventions: Other: exercise
- Uphill walking (Experimental): uphill walking training on the treadmill for 2 days/week
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — exercise training for 8 weeks

SUMMARY:
Selective exercise programs specific to muscle groups, with the workload to be done in line with the muscle's own structure, can enable more strength to be released with less fatigue in MS, and this increase in strength can increase balance and functional activities. to determine the effects of type training (selective exercise training), eccentric and concentric training on function, balance, fatigue and muscle architecture.

DETAILED DESCRIPTION:
Recovery and enhancement of muscle function in MS is one of the main goals in physiotherapy and rehabilitation. In literature studies, it is stated that eccentric and concentric exercises are effective exercise approaches in increasing strength and reducing fatigue. However, the best exercise method is not yet clear in terms of providing better performance adaptation with less fatigue. Considering the architectural features of the lower extremity muscles, it is aimed to increase the angle of pennation with programs that include concentric strengthening of the quadriceps, gastro-soleus and gastrocnemius muscles, which are suitable muscle groups to produce large forces by design. With programs that include eccentric strengthening of the hamstring and tibialis anterior muscles that function in a wide range of motion and have high excursion ability, it is aimed to increase fiber length.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-50,
* With an Extended Disability Status Scale (EDSS) score of 4 or less,
* No regular exercise habit
* Able to walk on the treadmill,
* No pregnancy,
* Not receiving corticosteroid treatment in the last month,
* Fampridine etc. in the last 1 month. not taking medication,
* Patients who have not received Botox treatment in the last 6 months

Exclusion Criteria:

patients who do not agree to volunteer

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
muscle architecture parameter 1 | Change from Baseline at 8th weeks and 12th weeks
  The pennation angle were evaluated with Ultrasound
muscle architecture parameter 2 | Change from Baseline at 8th weeks and 12th weeks
  The fiber length were evaluated with Ultrasound
muscle architecture parameter 3 | Change from Baseline at 8th weeks and 12th weeks
  The muscle thickness were evaluated with Ultrasound
Muscle strength | Change from Baseline at 8th weeks and 12th weeks
  low extremity muscles were evaluated with hand dynamometer

SECONDARY OUTCOMES:
walking fatigue | Change from Baseline at 8th weeks and 12th weeks
  Walking Fatigue Index
perceived fatigue | Change from Baseline at 8th weeks and 12th weeks
  Fatigue Severity Scale
physical fatigue | Change from Baseline at 8th weeks and 12th weeks
  Modified Borg Scale before and after 6-minute walking test
static balance | Change from Baseline at 8th weeks and 12th weeks
  Single standing tests
dynamic balance | Change from Baseline at 8th weeks and 12th weeks
  4 square step tests
Functional activities 1 | Change from Baseline at 8th weeks and 12th weeks
  timed-up go test
Functional activities 2 | Change from Baseline at 8th weeks and 12th weeks
  2-minute walk test
Functional activities 3 | Change from Baseline at 8th weeks and 12th weeks
  25-feet walk test

CONTACTS AND LOCATIONS:
Overall Officials: TÜZÜN FIRAT, Study Director — Hacettepe University; AYHAN ÖZKUR, Study Chair — Sanko University; AYŞE MÜNİFE NEYAL, Study Chair — Sanko University; ABDURRAHMAN NEYAL, Study Chair — Dr. Ersin Arslan Training and Research Hospital,; NEVİN ERGUN, Study Director — Sanko University
Locations (1):
- Zekiye İpek Katırcı Kırmacı, Gaziantep, Turkey (Türkiye)